CLINICAL TRIAL: NCT01767727
Title: Repair of Multiple Finger Defects Using the Dorsal Homodigital Island Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB-TS-0130067
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2012-10

CONDITIONS: Finger Injuries; Soft Tissue Injuries
Keywords: surgical flap;; dorsal branch of the digital artery
MeSH Terms: conditions — Finger Injuries; Soft Tissue Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical flap (Other): Surgical flap is based on the dorsal branch of the digital artery, and is used for soft tissue coverageof multiple finger defects.
  Interventions: Procedure: Soft tissue coverage

INTERVENTIONS:
Procedure: Soft tissue coverage — The dorsal homodigital island flaps are used for soft tissue coverage of multiple finger defects

SUMMARY:
Multiple finger defects are common in hand trauma and result in functional disability. These injuries are often complex and severe, and thus reconstructive alternatives are limited. In this study, we use the dorsal homodigital island flaps, based on the dorsal branch of the digital artery, for reconstruction of multiple finger defects. At the final follow-up, we would evaluate the efficacy of this technique.

DETAILED DESCRIPTION:
At final follow-up, sensation of the flap and the donor site would be assessed using static two-point discrimination and Semmes-Weinstein monofilament testing. The range of motion of the proximal interphalangeal joint and the distal interphalangeal joint of the injured finger is measured by a goniometer. The cold intolerance of the injured finger is measured using the self-administered Cold Intolerance Severity Score questionnaire that is rated into mild, moderate, severe, and extreme. The pain of the injured finger and the donor site is given subjectively by the patient using the visual analogue scale, which ranges from 0 to 10 cm and groupes into mild (0-3 cm), moderate (4-6 cm) and severe (7-10 cm).

ELIGIBILITY:
Inclusion Criteria:

1. a patient who had separate soft tissue defects in different fingers in same hand;
2. the defect ≥ 1.5 cm and ≤ 3.5 cm in length;
3. local tissue near the defect is uninjured; and
4. a patient between 15 and 60 years of age.

Exclusion Criteria:

1. concomitant injuries to local tissue around the defect that precluded its use as donor site;
2. a defect < 1.5 cm and ≥ 3.5 cm in length;
3. a finger degloving injury;
4. the defect of the thumb.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2011-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
static two-point discrimination | postoperative 18-24 months
  The test points are at the center of the flap.Each area is tested 3 times with a Discriminator. We stopp at 4 mm as a limit of two-point discrimination and consider this normal.

SECONDARY OUTCOMES:
Cold intolerance of the injured finger | Postoperative 18-24 months
  The cold intolerance of the injured finger was measured using the self-administered Cold Intolerance Severity Score questionnaire that was rated into mild, moderate, severe, and extreme.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Background] Hu HT, Chen WH, Liu WC, Hang QW. [Fingertip reconstruction using a volar flap based on the transverse palmar branch of the digital artery]. Zhonghua Zheng Xing Wai Ke Za Zhi. 2005 Sep;21(5):353-5. Chinese. PMID 16335381
- [Result] Al-Qattan MM. Technical modifications and extended applications of the distally based adipofascial flap for dorsal digital defects. Ann Plast Surg. 2004 Feb;52(2):168-73. doi: 10.1097/01.sap.0000101954.16674.99. PMID 14745267